CLINICAL TRIAL: NCT03721146
Title: ENCAPSID Study : Encapsulated Bacterial Infection and Primary, Secondary Immunodeficiency
Acronym: ENCAPSID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: RCB 2018-A00079-46
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-10

CONDITIONS: Immune Deficiency
Keywords: Encapsulated bacterial Infection; Primary immune deficiency; Secondary immune deficiency; Adult
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — complete blood count, blood smear, immunoglobulin (Ig) isotype (IgA,M, G) and IgG subclass levels, total hemolytic complement and complement fractions (C) 3 and 4, alternative complement pathway (AP50) in case of Neisseria meningitidis (NM) infection, quantitative immunophenotyping of T, B and natural killer cells, specific antibody response to diphtheria, tetanus and pneumococcal vaccine and HIV serology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background : The occurrence of Primary immune deficiencies (PID) is rare in adults. Antibody deficiencies were the first PID to be diagnosed in adulthood and are mainly represented by common variable immune deficiency. The main manifestation of these PID are encapsulated bacterial infection which used to be recurrent and/or invasive, lead to hospitalization and have high rates of morbidity and mortality. Diagnosis of PID in adulthood may be supported by six warning signs from the European Society of Immunodeficiencies (ESID). However, their guidelines do not comprehensively describe symptoms of PID, even for patients with infections. The guidelines recommend screening adults for PID after at least two severe bacterial infections. The aim of this study is to screen for PID adult admitted to our hospital for encapsulated infection without any predisposal factor.

Material and methods :

* Monocentric study. Inclusion between September 218 and September 2021
* Inclusion criteria :

  1. Age 18 to 65 years old
  2. Invasive encapsulated infection (Streptococcus pneumoniae, Streptococcus pyogènes, Haemophilus influenzae, Neisseiria meningitidis or Neisseria gonorrhoeae )
* Exclusion criteria :

  1. Medical history of PID
  2. Medical history of Secondary immune deficiency (SID)
  3. Local-regional factor that could predispose them to infection
  4. Hospital-acquired infection
* PID screening included the following: complete blood count, blood smear, immunoglobulin (Ig) isotype (IgA,M, G) and IgG subclass levels, total hemolytic complement and complement fractions (C) 3 and 4, alternative complement pathway (AP50) in case of Neisseria meningitidis (NM) infection, quantitative immunophenotyping of T, B and natural killer cells, specific antibody response to diphtheria, tetanus and pneumococcal vaccine and HIV serology. The clinical and laboratory diagnostic criteria used to identify PID were based on guidelines from the ESID and the Pan-American Group for Immunodeficiency (PAGID)
* A consultation in the infectious Diseases Department or Internal Medicine will be scheduled the hospitalization 3 months later to include patients and perform PID screening.

DETAILED DESCRIPTION:
Background : Primary immune deficiencies (PID) are characterized by a failure of the immune system that is not explained by any infectious, neoplastic, or iatrogenic causes. By 2017, more than 350 different inherited rare PID disorders had been described. The occurrence of PID is rare in adults, with a prevalence of approximately 6.7 per 100,000 inhabitants in France. Infections are the most common manifestations of PID .Theses Infections are usually recurrent and/or invasive, lead to hospitalization and have high rates of morbidity and mortality. Antibody deficiencies were the first PID to be diagnosed in adulthood and are mainly represented by common variable immune deficiency. The main manifestation of these PID are encapsulated bacterial infection. Diagnosis of PID in adulthood may be supported by six warning signs from the European Society of Immunodeficiencies (ESID). However, their guidelines do not comprehensively describe symptoms of PID, even for patients with infections. The guidelines recommend screening adults for PID after at least two severe bacterial infections. The aim of this study is to screen for PID adult admitted to our hospital for encapsulated infection without any predisposal factor.

Material and methods :

* Monocentric study. Inclusion between September 218 and September 2021
* Every months, micriobiologists will transfer to infectious diseases doctors and internal medicine doctors the name of patients who had a sample (cerebral fluid, articular fluid, blood culture, urine culture...) positive for Streptococcus pneumoniae, Streptococcus pyogenes, Haemophilus influenzae, Neisseiria meningitidis or Neisseria gonorrhoeae.
* Doctors will look at their medical records to see if they are eligible.
* Inclusion criteria :

  1. Age 18 to 65 years old
  2. Invasive encapsulated infection (Streptococcus pneumoniae, Streptococcus pyogènes, Haemophilus influenzae, Neisseiria meningitidis or Neisseria gonorrhoeae )
* Exclusion criteria :

  1. Medical history of PID
  2. Medical history of Secondary immune deficiency (SID)
  3. Local-regional factor that could predispose them to infection
  4. Hospital-acquired infection

     If patients are eligible, a consultation in the infectious Diseases Department or Internal Médicine Department will be scheduled the hospitalization 3 months later to include patients and perform PID screening.
* PID screening included the following: complete blood count, blood smear, immunoglobulin (Ig) isotype (IgA,M, G) and IgG subclass levels, total hemolytic complement and complement fractions (C) 3 and 4, alternative complement pathway (AP50) in case of Neisseria meningitidis (NM) infection, quantitative immunophenotyping of T, B and natural killer cells, specific antibody response to diphtheria, tetanus and pneumococcal vaccine and HIV serology. The clinical and laboratory diagnostic criteria used to identify PID were based on guidelines from the ESID and the Pan-American Group for Immunodeficiency (PAGID)

ELIGIBILITY:
Inclusion Criteria:

* Age :18 to 65 years old
* Admitted for an invasive encapsulated infection (Streptococcus pneumoniae, Streptococcus pyogènes, Haemophilus influenzae, Neisseiria meningitidis or Neisseria gonorrhoeae )

Exclusion criteria :

* Medical history of PID
* Medical history of Secondary immune deficiency (SID)
* A local-regional factor that could predispose them to infection (chronic pulmonary failure, cystic fibrosis, base scull fracture....)
* An hospital-acquired infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted for an invasive encapsulated infection without predisposing factors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients diagnosed for a primary immunodeficiency after admission for encapsulated bacterial infection | 3 months
  A consultation in the Internal Medicine or Infectious Diseases Department is scheduled 3 months after admission at the hospital for encapsulated bacterial infection to investigate an immune deficiency. This consultation consit on a physical examination and a immune testing. Immune testing included but is not limited to :
  Complete blood count, blood smear Immunoglobulin (Ig) isotype and IgG sub class quantitation (gram per litre) Quantitative serum complement (C3 (milligram per litre), C4 (milligram per litre), CH50 (%) and AP50 when Neisseria meningitides infection) Extensive immunophenotyping of T, B, and natural killer cells (cells/mm3) Specific antibody response to a variety of vaccine (milligram/litre) HIV serology. The outcome measure is the number of participants with abnormal laboratory or radiology values leading to primary immune deficiency diagnosis

SECONDARY OUTCOMES:
Number of patients diagnosed for a secondary immunodeficiency after admission for encapsulated bacterial infection | 3 months
  A consultation in the Internal Medicine or Infectious Diseases Department is scheduled 3 months after admission at the hospital for encapsulated bacterial infection to investigate an immune deficiency. This consultation consit on a physical examination and a immune testing. Immune testing included but is not limited to :
  Complete blood count, blood smear Immunoglobulin (Ig) isotype and IgG sub class quantitation (gram per litre) Quantitative serum complement (C3 (milligram per litre), C4 (milligram per litre), CH50 (%) and AP50 when Neisseria meningitides infection) Extensive immunophenotyping of T, B, and natural killer cells (cells/mm3) Specific antibody response to a variety of vaccine (milligram/litre) HIV serology. The outcome measure is the number of participants with abnormal laboratory or radiology values leading to secondary immune deficiency diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie BALDOLLI, MD, Principal Investigator — Infectious Diseases Department
Locations (1):
- Centre Hospitalier Universitaire Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conley ME, Notarangelo LD, Etzioni A. Diagnostic criteria for primary immunodeficiencies. Representing PAGID (Pan-American Group for Immunodeficiency) and ESID (European Society for Immunodeficiencies). Clin Immunol. 1999 Dec;93(3):190-7. doi: 10.1006/clim.1999.4799. No abstract available. PMID 10600329
- See also: French prevalence of primay immune deficiency — https://www.ceredih.fr
- See also: European Society for immunodeficiency and warning signs for primary immune deficency — https://esid.org